CLINICAL TRIAL: NCT04111874
Title: Parent-Led Cognitive-Behavioral Teletherapy for Anxiety in Youth With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric A Storch, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H45203
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Behavioral Therapy; Autism Spectrum Disorder; Anxiety Disorders; Obsessive-Compulsive Disorder; Social Anxiety Disorder; Generalized Anxiety Disorder; Specific Phobia
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Obsessive-Compulsive Disorder; Phobia, Social; Generalized Anxiety Disorder; Phobia, Specific

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Intensity Therapist Assistance (LTA) (Experimental): Parents will receive four 30-minute supportive video calls with a therapist over the 12 weeks of treatment.
  Interventions: Behavioral: Cognitive Behavioral Teletherapy LTA
- Standard Therapist Assistance (STA) (Active Comparator): Parents will receive ten 60-minute supportive video calls with a therapist over the 12 weeks of treatment.
  Interventions: Behavioral: Cognitive Behavioral Teletherapy STA

INTERVENTIONS:
Behavioral: Cognitive Behavioral Teletherapy LTA — Participating families will receive a copy of the book 'Helping Your Anxious Child, 2nd Edition', as well as the companion parent and child workbooks, to use at home and in session with the therapist. During each of the four videoconferencing sessions, therapists will serve to provide encouragement and support as the parent works through the program independently.
  Arms: Low-Intensity Therapist Assistance (LTA)
Behavioral: Cognitive Behavioral Teletherapy STA — Participating families will also receive a copy of the book 'Helping Your Anxious Child, 2nd Edition', as well as the companion parent and child workbooks, to use at home and in session with the therapist. During each of the ten videoconferencing sessions, therapists will guide the parent through the implementation of the program, including explaining materials, assisting to develop planned therapy activities with the child, and problem-solving as needed.
  Arms: Standard Therapist Assistance (STA)

SUMMARY:
This study implements an anxiety-focused, parent-led, therapist-assisted cognitive behavioral teletherapy for parents of youth with ASD and anxiety.

DETAILED DESCRIPTION:
Anxiety disorders affect 50-80% of children with autism spectrum disorder (ASD) and are associated with significant life impairment and worsening trajectory without treatment. The most effective psychotherapy for anxiety in youth with and without ASD is cognitive behavioral therapy (CBT), but many families are not able to access CBT due to the cost, practicalities of attending treatment sessions, and limited availability of trained therapists. Alternative models of service delivery are greatly needed, with particular promise of parent-led therapist-assisted (PLTA) models and telehealth delivery formats. Parents may benefit from additional information regarding how to optimize the delivery of CBT for youths with ASD given the potential impact of ASD symptomology on core CBT skills. Thus, this project aims to improve access to anxiety-focused Parent-Led Therapist-Assisted CBT for parents of youth with ASD. Parent-led low-intensity treatment models can improve accessibility, efficiency, and mental health treatment cost. Lower intensity treatment models provide a treatment option that is less costly and burdensome for parents; it is understood that some individuals will respond to the first step and others will require additional treatment to achieve anxiety reduction. However, understanding how many families, and which families, can benefit from a lower intensity model has dramatic benefits for improving access, allocating more intensive services for those most in need, and reducing barriers (e.g., distance). Thus, this study will examine the effectiveness of two anxiety-focused PTLA CBT telehealth models: 1) low-intensity therapist assistance (LTA) and 2) standard therapist assistance (STA). Overall, this study will provide important information regarding the potential benefits of two different approaches to parent-led interventions for youth with ASD and anxiety when delivered via telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Child is between the ages 7-13 years at consent/assent.
* The child meets criteria for ASD.
* The child meets criteria for clinically significant anxiety and/or OCD symptoms.
* Anxiety and/or OCD is the primary presenting problem.
* One parent/guardian is able and willing to participate.
* The child has a Full Scale and Verbal Comprehension Intelligence Quotient >70.
* The child is able to communicate verbally.
* Participants must reside in Texas and parents must be in the state of Texas when taking calls.

Exclusion Criteria:

* The child has a diagnosis of lifetime DSM-5 bipolar disorder, psychotic disorder, and/or intellectual disability.
* The child has severe current suicidal/homicidal ideation and/or self-injury requiring medical intervention.
* The child is receiving concurrent psychotherapy for anxiety.
* Initiation of a psychotropic medication less than 4 weeks prior to study enrollment or a stimulant/psychoactive medication less than 2 weeks prior to study enrollment.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guzick AG, Schneider SC, Kook M, Rose Iacono J, Weinzimmer SA, Quast T, Olsen SM, Hughes KR, Jellinek-Russo E, Garcia AP, Candelari A, Berry LN, Goin-Kochel RP, Goodman WK, Storch EA. Parent-Led Cognitive Behavioral Teletherapy for Anxiety in Autistic Youth: A Randomized Trial Comparing Two Levels of Therapist Support. Behav Ther. 2024 May;55(3):499-512. doi: 10.1016/j.beth.2023.08.008. Epub 2023 Sep 6. PMID 38670664
- [Derived] Greenberg RL, Guzick AG, Schneider SC, Weinzimmer SA, Kook M, Perozo Garcia AB, Storch EA. Depressive Symptoms in Autistic Youth with Anxiety Disorders. J Dev Behav Pediatr. 2023 Dec 1;44(9):e597-e603. doi: 10.1097/DBP.0000000000001223. Epub 2023 Oct 11. PMID 38019467
- [Derived] Elliott SJ, Marshall D, Morley K, Uphoff E, Kumar M, Meader N. Behavioural and cognitive behavioural therapy for obsessive compulsive disorder (OCD) in individuals with autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2021 Sep 3;9(9):CD013173. doi: 10.1002/14651858.CD013173.pub2. PMID 34693989

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-Intensity Therapist Assistance (LTA) | Standard Therapist Assistance (STA)
Started | 48 | 39
Completed | 31 | 35
Not Completed | 17 | 4

BASELINE CHARACTERISTICS:
Population: All participants (87) were randomly assigned to either the LTA or STA groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Intensity Therapist Assistance (LTA) | Standard Therapist Assistance (STA) | Total
Number analyzed (Participants) | 48 | 39 | 87
Age, Categorical [Count of Participants; unit: Participants] — Population: Individuals were randomly assigned to different conditions
  Participants
    <=18 years | 48 | 39 | 87
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants were randomly assigned to different conditions
  years | 10.1 (1.8) | 10.3 (1.8) | 10.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants were randomly assigned to different conditions
  Participants
    number analyzed (Participants) | 46 | 38 | 84
    Female | 8 | 8 | 16
    Male | 38 | 30 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants were randomly assigned to different conditions
  Participants
    Hispanic or Latino | 17 | 11 | 28
    Not Hispanic or Latino | 29 | 27 | 56
    Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants were randomly assigned to different conditions
  Participants
    American Indian or Alaska Native | 1 | 2 | 3
    Asian | 3 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 2 | 4
    White | 33 | 23 | 56
    More than one race | 7 | 11 | 18
    Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants] — Population: Participants were randomly assigned to different conditions
  participants
    United States | 48 | 39 | 87

OUTCOME MEASURES:

1. Primary Outcome: 6-item Pediatric Anxiety Rating Scale
Description: Clinician rated child anxiety severity throughout the past week. Each item is scored on a 0 to 5 scale (higher scores correspond to greater severity), yielding a total between 0 and 30.
Time Frame: Baseline (before treatment), post-treatment (on average 12 weeks), 3 month follow up; Post-treatment scores reported.
Population: Results for the post-treatment assessment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Low-Intensity Therapist Assistance (LTA) | Standard Therapist Assistance (STA)
Number analyzed (Participants) | 31 | 33
Score on a scale | 11.35 (5.36) | 10.26 (4.17)

2. Primary Outcome: Clinical Global Impression-Improvement
Description: Clinician rated child psychopathology improvement since initial rating. A single item is scored 0-6 (0 = very much worse; 6= very much improved).
Time Frame: Each treatment session, post-treatment (on average 12 weeks), 3 month follow up; Post-treatment scores reported.
Population: count of participants who were classified as "much" or "very much improved" on the CGI-I at the end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Intensity Therapist Assistance (LTA) | Standard Therapist Assistance (STA)
Number analyzed (Participants) | 31 | 33
Participants | 21 | 23

3. Secondary Outcome: Clinical Global Impression-Severity
Description: Clinician rated child psychopathology severity rating. A single item is scored 0-6 (0= no illness; 6= extremely severe symptoms).
Time Frame: Baseline (before treatment), Each treatment session, post-treatment (on average 12 weeks), 3 month follow up; Post-treatment scores reported.
Population: These scores are reported for the post-treatment assessment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Low-Intensity Therapist Assistance (LTA) | Standard Therapist Assistance (STA)
Number analyzed (Participants) | 31 | 33
Score on a scale | 2.83 (1.07) | 2.59 (1.08)

ADVERSE EVENTS:
Time Frame: Participants were enrolled in the study for up to 6 months, which corresponds to the time that adverse event data were collected
Description: Definition of adverse event does not differ from that of clinicaltrails.gov
Arm/Group | Low-Intensity Therapist Assistance (LTA) | Standard Therapist Assistance (STA)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/39
Other Adverse Events (participants affected / at risk) | 0/48 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-08-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT04111874/Prot_SAP_ICF_000.pdf